CLINICAL TRIAL: NCT04321018
Title: Effect of the Addition of Medium Chain Triglycerides to a Mixed Macronutritional Meal on the Oxidation of Postprandial Macronutrients
Brief Title: Effect of a Mixed Macronutritional Meal With Medium Chain Triglycerides on the Oxidation of Postprandial Macronutrients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Associate professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: nº 1102/CEIH/2020
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal with medium chain triglycerdies first (Experimental): Arm 1: participants randomized to receive the mixed meal with medium chain triglycerides first.
  Interventions: Dietary Supplement: Mixed meal with medium chain triglycerides; Dietary Supplement: Mixed meal with the replacement of medium chain triglycerides with unsaturated tryglicerides
- Meal with medium chain triglycerdies second (Active Comparator): Arm 2: participants randomized to receive the mixed meal without medium chain triglycerides first.te
  Interventions: Dietary Supplement: Mixed meal with medium chain triglycerides; Dietary Supplement: Mixed meal with the replacement of medium chain triglycerides with unsaturated tryglicerides

INTERVENTIONS:
Dietary Supplement: Mixed meal with medium chain triglycerides — Mixed macronutrient liquid meal (1.6kcal/ml, 15% protein, 47% carbohydrates, 35% fat, 3% fiber) with medium chain triglycerides (3g/100 kcal). An amount with energy supply equivalent to their 50% basal metabolic rate.
Dietary Supplement: Mixed meal with the replacement of medium chain triglycerides with unsaturated tryglicerides — Mixed macronutrient liquid meal (1.6kcal/ml, 15% protein, 47% carbohydrates, 35% fat, 3% fiber) without medium chain triglycerides (replaced it with long chain triglycerides). An amount with energy supply equivalent to their 50% basal metabolic rate.

SUMMARY:
The main aim of this study is to determine the effect of the addition of medium chain triglycerides to a mixed macro nutritional meal on postprandial macronutrients oxidation (i.e. fat oxidation, carbohydrate oxidation, change in respiratory quotient, peak respiratory quotient, etc.).

DETAILED DESCRIPTION:
A mixed meal characterized by a high quantity of carbohydrates could develop an increment in the postprandial carbohydrate oxidation. Medium chain triglycerides could be absorbed and metabolized immediately. It is plausible that its addition to a mixed meal unchains the decrement in the carbohydrate oxidation and increment in fat oxidation. If this hypothesis it is correct, its lower postprandial carbohydrate oxidation could develop a higher postprandial exposure to hyperglycemia, being of clinical interest.

20 young adults will be randomized into two conditions (experimental and control conditions) with 7 days of separation between conditions. Each evaluation day will conform to the following tests:

1. Basal metabolic rate assessment through indirect calorimetry.
2. Intake of the corresponding mixed meal (experimental or control)
3. Postprandial nutrient oxidation and energy expenditure through indirect calorimetry
4. Blood samples assessment in 9 time points during the evaluation day.
5. Post-prandial sensations related to appetite in 11 time points during the evaluation day

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Ages 18-30 years
* BMI: 18-27.5 kg/m2
* Stable weight over the last 3 months (body weight changes<35kg)
* Participant must be capable and willing to provide consent, understand exclusion criteria, instructions and protocols.

Exclusion Criteria:

* History of cardiovascular disease
* Diabetes or hypertension
* Pregnant, planning to become pregnant, or breastfeeding
* Have been treated previously or during the study period with prescription drugs: antihypertensive, lipid lowering, acid uric lowering, glucose lowering, beta blockers or any drug that under the investigator's judged could influence the results.
* Hematological pathology
* Have had a blood transfusion or severe blood loss within the last 3 months
* Allergy/intolerance to milk proteins, fish, soy, and/or any ingredient of the mixed meal
* Any non-controlled medical condition which could influence results or could be worsened by the participation in the study
* Claustrophobia
* Needle phobia
* Are deemed unsuitable by the investigator for any other reason, that prevent data collection.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Post-prandial nutrient oxidation | 4 hours
  Fat or carbohydrate oxidation measured by indrect calorimetry

SECONDARY OUTCOMES:
Post-prandial blood glucose concentrations | 4 hours
  Measures of blood glucose concentrations
Post-prandial blood insulin concentrations | 4 hours
  Measures of blood insulin concentrations
Post-prandial blood non-esterified fatty acid concentrations | 4 hours
  Measures of blood non-esterified fatty acid concentrations
Post-prandial blood tryglicerides concentrations | 4 hours
  Measures of blood tryglicerides concentrations
Post-prandial blood cholesterol concentrations | 4 hours
  Measures of blood cholesterol concentrations
Post-prandial blood glycerol concentrations | 4 hours
  Measures of blood glycerol concentrations
Post-prandial blood lactate concentrations | 4 hours
  Measures of blood lactate concentrations
Post-prandial energy expenditure | 4 hours
  Measured by indrect calorimetry
Post-prandial sensations related to appetite | 4 hours
  Measured by visual analogue scales (VAS). Score ranging from 0 to 100mm. Higher values mean the most positive rating, while lower values mean the most negative rating.

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan Ruiz Ruiz, Dr., Principal Investigator — Universidad de Granada
Locations (1):
- Jonatan Ruiz Ruiz, Granada, Spain

IPD SHARING:
Plan to Share IPD: No